CLINICAL TRIAL: NCT06804434
Title: Impact of Intraoperative Non-invasive Analgesia Monitoring Using Nociception Level Index on Patient Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osoian Cristiana (Other)
Responsible Party: Sponsor-Investigator, Osoian Cristiana, Principal Investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Organization: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: NOL-1047
Record Dates: First submitted 2025-01-19; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pain; Anesthesia; Perioperative Care
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- + NOL + lidocaine group (Experimental): NOL guided analgesia and intravenous lidocaine infusion
  Interventions: Drug: Lidocaine Intravenous Infusion; Device: NOL
- - NOL - lidocaine group (No Intervention): group without NOL monitoring or lidocaine administration
- + NOL - lidocaine group (Experimental): NOL guided analgesia without intravenous lidocaine infusion
  Interventions: Device: NOL
- - NOL + lidocaine group (Experimental): group without NOL monitoring but with lidocaine intravenous infusion
  Interventions: Drug: Lidocaine Intravenous Infusion

INTERVENTIONS:
Drug: Lidocaine Intravenous Infusion — intravenous lidocaine 10 mg/ml continuous infusion
  Arms: + NOL + lidocaine group; - NOL + lidocaine group
Device: NOL — Intraoperative Nociception Level index monitoring and guided analgesia
  Arms: + NOL + lidocaine group; + NOL - lidocaine group

SUMMARY:
This prospective randomised clinical trial aims to assess the impact of intraoperative nociception monitoring using NOL on anesthetic management during major abdominal surgery. Additionally, the study will objectively evaluate using NOL how intravenous lidocaine administration, influences opioid requirements and the effect of this multimodal approach on early postoperative outcomes. The investigators hypothesize that NOL-guided intraoperative opioid administration reduces both intraoperative and postoperative opioid use, positively influencing 24-hour outcomes. Furthermore, the addition of intraoperative lidocaine in NOL-guided analgesia may further decrease opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* ASA score I-III
* surgery for gastric or hepatobiliary or pancreatic neoplasia

Exclusion Criteria:

* pregnancy
* lactation
* neuraxial or regional anesthesia
* chronic treatment with drugs that can influence autonomic nervous system
* diuretics or nitroglycerin administration on the day of surgery
* severe neurological disability
* severe hemodynamic instability
* chronic pain
* chronic opioid treatment
* allergy to any of the study drugs
* severe untreated disease or organ failure
* pacemaker
* emergency surgery
* patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative opioid use | intraoperative
  We aim to examine the effect nociception level index monitoring in major abdominal surgery on intraoperative nociception management by measuring total opioid use in NOL monitored patients vs standard care according to the anesthesiologists judgement. Moreover, crossreference interventional arms will examine the effect of intraoperative administration of lidocaine in NOL and no NOL groups on intraoperative opioid use. Intraoperative opioid use will be time adjusted ( depending on the duration of surgery) and weight adjusted (depending on the weight of the patient)- mg of opioid/hour/kg

SECONDARY OUTCOMES:
Intraoperative pulse | intraoperative
  Mean pulse rate and peak pulse rate
Intraoperative blood pressure | intraoperative
  Mean blood pressure and peak blood pressure
Postoperative pain scores | 24 hours
  VAS score at 15 minutes, 30 minute, 2 hours 4 hours, 12 hours and 24 hours
Postoperative opioid use | 24 hours
Lidocaine related adverse events | 24 hours
Opioid related adverse events | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Gastroenterology and Hepatology Institute Octavian Fodor, Cluj-Napoca, Cluj, Romania